CLINICAL TRIAL: NCT04663984
Title: Publication Rates of Theses in the Field of Anesthesiology and Reanimation in Turkey; Analysis of 2563 Theses
Brief Title: Analysis of 2560 Theses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, İLKE KÜPELİ, assoc. prof., Derince Training and Research Hospital
Other Study IDs: derince TRH 1
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Publication Rates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: publication rates — publication rates of theses produced in the Department of Anesthesiology and reanimation

SUMMARY:
Thesis publication rates in our country, according to research other medical branches; in psychiatry thesis % 37,4; Family Medicine, an increase of 0.9%; in emergency medicine and 7.3% in public health 1.5%; in microbiology %4,2; 5.7 percent in urology; brain surgery was 6.8%; general surgery 5%; 3.8% in eye diseases and surgery; ear, nose and throat diseases and surgery, in %4,2 as has been reported.

ELIGIBILITY:
Inclusion Criteria:

* the keywords" anesthesiology and reanimation"
* Made between 2000 and 2018,
* theses whose complete data can be accessed and allowed to be accessed by authors over the internet

Exclusion Criteria:

* theses whose complete data can be accessed and whose access is not allowed by the authors over the internet.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 2563 theses made between 2000 and 2018 using the keywords" anesthesiology and reanimation", full data of which can be accessed and allowed to be accessed by the authors over the internet.
Sampling Method: Non-Probability Sample
Enrollment: 2563 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
publication rate | 2 month
  publication rates of theses produced in the Department of Anesthesiology and reanimation

CONTACTS AND LOCATIONS:
Locations (1):
- derince TRH, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Erim BR, Petekkaya S. Retrospective Analysis of Psychiatry Specialization Theses Made Between 1981-2018 in Turkey. Turk Psikiyatri Derg. 2020 Spring;31(1):1-8. doi: 10.5080/u23877. English, Turkish. PMID 32594474
- [Result] Sipahi OR, Caglayan Serin D, Pullukcu H, Tasbakan M, Koseli Ulu D, Yamazhan T, Arda B, Sipahi H, Ulusoy S. [Publication rates of Turkish medical specialty and doctorate theses on Medical Microbiology, Clinical Microbiology and Infectious Diseases disciplines in international journals]. Mikrobiyol Bul. 2014 Apr;48(2):341-5. doi: 10.5578/mb.7003. Turkish. PMID 24819272